CLINICAL TRIAL: NCT01313988
Title: Efficacy Study on the Lipid-lowering Effect of a Spread Enriched With the Recommended Dose of Plant Sterols and 3 Different Doses of Fatty Acids From Fish Oil
Brief Title: Efficacy Study on the Lipid-lowering Effect of Plant Sterols and Fish Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10018V
Record Dates: First submitted 2011-03-02; First posted 2011-03-14 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Healthy; Mildly Elevated Cholesterol Levels
Keywords: dose-response study; blood lipid profile; plant sterols; fish oil
MeSH Terms: interventions — Phytosterols; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose 1 (Active Comparator): Spread that contains plant sterols and fish oil
  Interventions: Dietary Supplement: Plant sterols and fish oil
- Dose 2 (Active Comparator): Spread that contains plant sterols and fish oil
  Interventions: Dietary Supplement: Plant sterols and fish oil
- Dose 3 (Active Comparator): Spread that contains plant sterols and fish oil
  Interventions: Dietary Supplement: Plant sterols and fish oil
- Placebo (Placebo Comparator): Placebo spread
  Interventions: Dietary Supplement: Placebo
- Control (Active Comparator): Spread that contains plant sterols
  Interventions: Dietary Supplement: Plant sterols

INTERVENTIONS:
Dietary Supplement: Plant sterols and fish oil — 4 weeks intervention, 3 times daily
  Arms: Dose 1; Dose 2; Dose 3
Dietary Supplement: Plant sterols — 4 weeks intervention, 3 times daily
  Arms: Control
Dietary Supplement: Placebo — 4 weeks, 3 times daily
  Arms: Placebo

SUMMARY:
Plant sterols and fish fatty acids are known to affect the blood lipid profile. This randomized, double-blind, placebo-controlled, parallel efficacy study is designed to investigate the lipid-lowering effect after 4 weeks intervention with the recommended dose of plant sterols and different doses of fish fatty acids when combined in a spread format.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women
* Age ≥ 25 and ≤ 75 years old
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2
* Total cholesterol levels at screening ≥ 5.0 and ≤ 8.0 mmol/L
* 10-year CVD risk equal or lower than 10% according to "SCORE"
* Blood pressure, heart rate, hematological parameters, clinical chemical parameters within normal reference ranges
* Informed consent and biobank consent signed
* Willing to comply to study protocol during study
* Agreeing to be informed about medically relevant personal test-results by a physician
* Not smoking
* Accessible veins on the forearm
* Habitually consuming spreads

Exclusion Criteria:

* Pregnant or having the wish to become pregnant, or lactating
* Use of prescribed medication which may interfere with study measurements
* Use of antibiotics in the 3 months before screening or during the study
* Use of any medically- or self-prescribed diet with the purpose to reduce weight
* Intolerance for gluten or lactose
* Reported food allergy
* Having bleeding disorders
* Recent blood donation
* Excessive alcohol consumption
* Strenuous exercise
* Reported weight change ≥ 10 % of body weight or use of prescribed weight reduction drugs
* Recent participation in another nutritional or medical trial
* Participation in night shift work

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in blood lipid profile | At baseline (after 4 weeks run-in period) and after 4 weeks intervention
  Includes total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides

SECONDARY OUTCOMES:
Change in EPA/DHA in red blood cells | At baseline (after 4 weeks run-in period) and after 4 weeks intervention
Change in metabolomic parameters | At baseline (after 4 weeks run-in period) and after 4 weeks intervention
  For exploratory purposes

CONTACTS AND LOCATIONS:
Overall Officials: Johan Olsson, PhD, Principal Investigator — KPL Good Food Practice AB; Birgitta Sundberg, PhD, Study Director — KPL Good Food Practice AB; Anneli Hallmin, Study Director — KPL Good Food Practice AB
Locations (1):
- KPL Good Food Practice AB, Uppsala, Sweden

REFERENCES:
- [Derived] Ras RT, Demonty I, Zebregs YE, Quadt JF, Olsson J, Trautwein EA. Low doses of eicosapentaenoic acid and docosahexaenoic acid from fish oil dose-dependently decrease serum triglyceride concentrations in the presence of plant sterols in hypercholesterolemic men and women. J Nutr. 2014 Oct;144(10):1564-70. doi: 10.3945/jn.114.192229. Epub 2014 Aug 13. PMID 25122648